CLINICAL TRIAL: NCT01933555
Title: Impact of Women's Empowerment Program for Abused Pregnant Women: A Randomized Controlled Trial
Brief Title: Impact of Women's Empowerment Program for Abused Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Macmillan Research Group UK (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mac/NMP 0912
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Abuse Physical Battered Woman Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Empowerment program (Experimental): The hour intervention, delivered over a 11-week period, consisted of an empowerment and additional components adapted from Freedom program run to support domestic abused women.
  Interventions: Behavioral: Empowerment Program
- Control group (No Intervention): Standard care, which was routine check ups and care provided by health care professionals.

INTERVENTIONS:
Behavioral: Empowerment Program
  Arms: Empowerment program

SUMMARY:
Although domestic violence is recognized as major threat in pregnancy, there is no intervention has been developed or test to support women in India. To evaluate the effect of women's empowerment program administered to abused women in order to reduce domestic abuse, improving health status and safety behavior.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age,
* victims of intimate partner violence, and
* willing to participate

Exclusion Criteria:

* women whose abuser was not their intimate partner or
* who were unable to consent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Quality of life(Sf-36) | Five Months

SECONDARY OUTCOMES:
Post natal depression | 5 months

OTHER OUTCOMES:
Domestic Violence Inventory and safety seeking behavior | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Macmillan research group
Locations (1):
- NMP medical research institute, Jaipur, Rajasthan, India